CLINICAL TRIAL: NCT00684086
Title: English Diabetes Self-Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 96943; 5312
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2008-05-26 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Behavioral: Diabetes Self Management Program

SUMMARY:
We propose a diabetes self-management program evaluation and dissemination project with three components.

1. A six-month randomized trial to evaluate the effect of a community-based small group Diabetes Self Management Program (DSMP) on the health related quality of life, metabolic control and health care utilization of people with type 2 diabetes.
2. A long-term (12 month) longitudinal evaluation of the same program.
3. Two 5 day workshops to train others in California in how to lead and administer the program.

DETAILED DESCRIPTION:
1. Implement and evaluate in a 6-month randomized controlled evaluation an experimental self-management program for patients with type 2 diabetes. Outcomes for evaluating the intervention's impact include health status (health-related quality-of-life and metabolic control) and health care utilization. Mediating outcomes are health behaviors and self-efficacy.
2. Evaluate the same program in a one year longitudinal study using the same outcomes.
3. Disseminate the program to others in California by holding two five day workshops during which we will prepare the participants to both offer the program and to train others in their organization to offer the program.

This proposed evaluation will examine the following questions:

Hypothesis 1. People participating in the Diabetes Self-Management Program (SDSMP), when compared six months after baseline to randomized wait-list controls receiving usual care, will demonstrate:

1. Improvements in health-related quality of life (fatigue, physical discomfort, the symptoms of hypoglycemia and hyperglycemia, activity limitations, health distress, and self-rated health).

   Improvements in metabolic measures of health status (body mass index, hemoglobin A1c, total cholesterol/HDL ratio and blood pressure).
2. Changes in utilization of health services, specifically, increases in outpatient visits to physicians and nurses, increases in the percentage of subjects having received an eye examination in the past year, increases in the number of times a health professional has examined subject's feet, and decreases in emergency room visits, hospitalizations, and hospital days.
3. Improvements in beneficial self-management behaviors (aerobic exercise, communication with physicians, diet, self-monitoring of blood glucose and self-examination of the feet).
4. Increases in perceived self-efficacy to manage diabetes.

Hypothesis 2. The changes in health related quality of life, metabolic status, health behaviors and health care utilization will be maintained for one year.

Hypothesis 3. Twelve to fifteen health care organizations in California will be interested in disseminating the program. This will be demonstrated by their willingness to send 2-3 persons each to a 5 day training which will allow their organization to replicate and perpetuate the program.

Hypothesis 4. 8-10 health care organizations in California will have offered at least two Diabetes Self-Management Programs to people with Type 2 diabetes one year following the above dissemination training. (It should be noted that this hypothesis can not be tested during the funded portion of the program. However, it our intent to contact all organizations participating in dissemination training one year following the training to determine what they have done with the program). The results of this follow-up will be reported to The Foundation.)

ELIGIBILITY:
Inclusion Criteria:

* Individuals with prior diagnosis of type 2 Diabetes.
* Able to speak and comprehend English.
* Able to give and complete consent forms.
* Able to complete baseline questionnaire and 2-3 follow-up questionnaires either in writing or by telephone.
* Able to attend respective community meetings or allow study staff to collect the following metabolic test measures: provide 3 drops of blood for Hemoglobin A1c and cholesterol HDL test (administered by subject), blood pressure measure, height and weight measures.
* Able to attend the Peer-Led Community-Based Diabetes Self-Management Program workshops offered once a week for six weeks at a community site near subjects residence.

Exclusion Criteria:

* Individuals not diagnosed with type 2 diabetes.
* Individuals diagnosed with type 1 diabetes.
* Pregnant women, including those diagnosed with gestational diabetes.
* Individuals who have been in active treatment for cancer in the past yar.
* Individuals not able to speak or comprehend English.
* Individuals who are currently or have previously participated in a similar program or study.
* Individuals that are not able to give consent or complete consent forms, and other study related forms such as questionnaires.
* Individuals who are not able and willing to provide metabolic test data.
* Individuals not able to attend the 6-week community classes in the target counties in California.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2007-04

PRIMARY OUTCOMES:
hemoglobin A1
symptoms of hypoglycemia
symptoms of hyperglycemia
self-monitoring of blood glucose
self-efficacy to manage diabetes

SECONDARY OUTCOMES:
fatigue
physical discomfort
activity limitations
health distress
self-rated health
aerobic exercise
communication with physicians

CONTACTS AND LOCATIONS:
Overall Officials: Kate R Lorig, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Lorig K, Ritter PL, Villa FJ, Armas J. Community-based peer-led diabetes self-management: a randomized trial. Diabetes Educ. 2009 Jul-Aug;35(4):641-51. doi: 10.1177/0145721709335006. Epub 2009 Apr 30. PMID 19407333